CLINICAL TRIAL: NCT02667821
Title: Changes in Vertebral Artery and Cerebral Hemodynamics Following Various Head Positions & Cervical Manipulation in Patients With Chronic/Recurrent Neck Pain
Brief Title: Vertebral Artery and Cerebral Hemodynamics After Various Head Positions & Manipulation in Patients With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Memorial Chiropractic College (Other)
Collaborators: National Chiropractic Mutual Insurance Company (NCMIC) (Unknown)
Responsible Party: Principal Investigator, Nick Moser, Local contact investigator, Canadian Memorial Chiropractic College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 162001
Record Dates: First submitted 2016-01-18; First posted 2016-01-29 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-09

CONDITIONS: Vertebral Artery Dissection; Cerebrovascular Accident; Stroke
MeSH Terms: conditions — Vertebral Artery Dissection; Stroke | interventions — Manipulation, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Experimental): Participants included in the experimental arm will be adults aged 18 years and older with chronic/recurrent neck pain Grade II who have been prescribed cervical manipulation for treatment of their condition. Each participant will undergo three separate test maneuvers consistent with prior work completed at the St. Joseph's Healthcare Hamilton Brain Body Institute. Each participant will begin with neutral cervical spine as a standard natural control, followed by block randomization between maximum voluntary rotation of the cervical spine and one cervical manipulation. Please see Intervention section for a detailed description.
  Interventions: Other: Head positions and spinal manipulation

INTERVENTIONS:
Other: Head positions and spinal manipulation — Each participant will undergo three separate test maneuvers. Neutral (0° rotation) neck position (condition 1) will be followed by block randomization between maximum voluntary rotation (condition 2) and a high-velocity-low-amplitude cervical manipulation targeted at C1-C2 (condition 3). Conditions 1 and 2 will be held for 1 minute before returning to neutral alignment. For the manipulation, the head will be repositioned at neutrality immediate. An experienced practitioner will perform the manipulation on the adjustable and pivotal MRI bed. After each condition, MRI of the upper neck and cerebrum for perfusion and blood flow will ensue.

SUMMARY:
The Investigators are performing a study to determine, in patients with chronic/recurrent neck pain, the cerebrovascular hemodynamic consequences of cervical spine movements, including manipulation, in vivo using fMRI technology on vertebral and cranial blood flow dynamics affecting brain perfusion, and extend the current data set on these variables

DETAILED DESCRIPTION:
The goal of the study is to further investigate in patients with chronic/recurrent neck pain, the cerebrovascular hemodynamic consequences of cervical spine positions, including manipulation, in vivo under clinically relevant circumstances using two advanced MRI technology on the vertebral and posterior cerebral and cerebellar blood flow dynamics affecting brain perfusion. According to the knowledge of the investigators, a study utilizing MRI to examine blood flow and perfusion, turbulence and evidence of micro-trauma within these blood vessels has yet to be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older with chronic/recurrent neck pain Grade II.
2. Must have been prescribed cervical spinal manipulation for treatment of their neck pain condition.

Exclusion Criteria:

1. A history of neck pain with associated arm pain within the last 6 months
2. Any current or history of neurologic symptoms including facial or extremity weakness, abnormal sensation to the face, body, or extremities, uncontrolled movements, abnormal gait, dizziness, unexplained nausea/vomiting, difficulty with speaking or swallowing
3. History of new or severe (Visual Analogue Scale >6) headaches in the last 3 months
4. Any contraindications to MRI
5. Any history of using drugs that affect blood flow such as Warfarin, or anti-coagulants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Wells, PhD, Principal Investigator — University of Toronto; Nicholas Moser, BSc, Dc, Principal Investigator — Canadian Memorial Chiropractic College; John J Triano, DC, PhD, Study Chair — Canadian Memorial Chiropractic College; Michael Noseworthy, PhD, Study Director — McMaster University; Silvano Mior, DC, PhD, Principal Investigator — Canadian Memorial Chiropractic College
Locations (1):
- St. Joseph Healthcare, Research Imaging Institute, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Study results will be made public through peer-reviewed journal publications, presentations, clinical trial registration and report to participants. If participants are interested in information on the outcome of the study they may request a report from their own data and / or aggregated data either at the time of consent and data capture by signing an area on the informed consent document or subsequently by written request to the principal investigator. ROF will be submitted to indexed and peer-reviewed journals interested in imaging and clinical biomechanics of the spine.

REFERENCES:
- [Background] Boyle E, Cote P, Grier AR, Cassidy JD. Examining vertebrobasilar artery stroke in two Canadian provinces. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S194-200. doi: 10.1016/j.jmpt.2008.11.019. PMID 19251064
- [Background] Cassidy JD, Boyle E, Cote P, He Y, Hogg-Johnson S, Silver FL, Bondy SJ. Risk of vertebrobasilar stroke and chiropractic care: results of a population-based case-control and case-crossover study. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S201-8. doi: 10.1016/j.jmpt.2008.11.020. PMID 19251066
- [Background] Rubinstein SM, Peerdeman SM, van Tulder MW, Riphagen I, Haldeman S. A systematic review of the risk factors for cervical artery dissection. Stroke. 2005 Jul;36(7):1575-80. doi: 10.1161/01.STR.0000169919.73219.30. Epub 2005 Jun 2. PMID 15933263
- [Background] Zaina C, Grant R, Johnson C, Dansie B, Taylor J, Spyropolous P. The effect of cervical rotation on blood flow in the contralateral vertebral artery. Man Ther. 2003 May;8(2):103-9. doi: 10.1016/s1356-689x(02)00155-8. PMID 12890438
- [Background] Cagnie B, Jacobs F, Barbaix E, Vinck E, Dierckx R, Cambier D. Changes in cerebellar blood flow after manipulation of the cervical spine using Technetium 99m-ethyl cysteinate dimer. J Manipulative Physiol Ther. 2005 Feb;28(2):103-7. doi: 10.1016/j.jmpt.2005.01.005. PMID 15800509
- [Background] Mitchell JA. Changes in vertebral artery blood flow following normal rotation of the cervical spine. J Manipulative Physiol Ther. 2003 Jul-Aug;26(6):347-51. doi: 10.1016/S0161-4754(03)00074-5. PMID 12902962
- [Background] Johnson C, Grant R, Dansie B, Taylor J, Spyropolous P. Measurement of blood flow in the vertebral artery using colour duplex Doppler ultrasound: establishment of the reliability of selected parameters. Man Ther. 2000 Feb;5(1):21-9. doi: 10.1054/math.1999.0227. PMID 10688956
- [Background] Sakaguchi M, Kitagawa K, Hougaku H, Hashimoto H, Nagai Y, Yamagami H, Ohtsuki T, Oku N, Hashikawa K, Matsushita K, Matsumoto M, Hori M. Mechanical compression of the extracranial vertebral artery during neck rotation. Neurology. 2003 Sep 23;61(6):845-7. doi: 10.1212/01.wnl.0000078081.12097.ae. PMID 14504337
- [Background] Haynes MJ. Doppler studies comparing the effects of cervical rotation and lateral flexion on vertebral artery blood flow. J Manipulative Physiol Ther. 1996 Jul-Aug;19(6):378-84. PMID 8864968
- [Background] Licht PB, Christensen HW, Hojgaard P, Hoilund-Carlsen PF. Triplex ultrasound of vertebral artery flow during cervical rotation. J Manipulative Physiol Ther. 1998 Jan;21(1):27-31. PMID 9467098
- [Background] Licht PB, Christensen HW, Svendensen P, Hoilund-Carlsen PF. Vertebral artery flow and cervical manipulation: an experimental study. J Manipulative Physiol Ther. 1999 Sep;22(7):431-5. doi: 10.1016/s0161-4754(99)70030-8. PMID 10519558
- [Background] Bendick PJ, Jackson VP. Evaluation of the vertebral arteries with duplex sonography. J Vasc Surg. 1986 Mar;3(3):523-30. doi: 10.1067/mva.1986.avs0030523. PMID 3512861
- [Derived] Moser N, Mior S, Noseworthy M, Cote P, Wells G, Behr M, Triano J. Effect of cervical manipulation on vertebral artery and cerebral haemodynamics in patients with chronic neck pain: a crossover randomised controlled trial. BMJ Open. 2019 May 28;9(5):e025219. doi: 10.1136/bmjopen-2018-025219. PMID 31142519

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty patients were recruited from the campus-teaching clinic located at the Canadian Memorial Chiropractic College. Included were adults aged 18 years and older with chronic grade II mechanical neck pain that had been prescribed cervical manipulation for treatment of their condition
Groups:
- Intervention Group: Participants included in the experimental arm will be adults aged 18 years and older with chronic/recurrent neck pain Grade II who have been prescribed cervical manipulation for treatment of their condition. Each participant will undergo three separate test maneuvers. Neutral (0° rotation) neck position (condition 1) will be followed by block randomization between maximum voluntary rotation (condition 2) and a high-velocity-low-amplitude cervical manipulation targeted at C1-C2 (condition 3). Conditions 1 and 2 will be held for 1 minute before returning to neutral alignment. For the manipulation, the head will be repositioned at neutrality immediate. An experienced practitioner will perform the manipulation on the adjustable and pivotal MRI bed. After each condition, MRI of the upper neck and cerebrum for perfusion and blood flow will ensue.
Period: Overall Study
Arm/Group | Intervention Group
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Each participant will undergo three separate test maneuvers. Neutral (0° rotation) neck position (condition 1) will be followed by block randomization between maximum voluntary rotation (condition 2) and a high-velocity-low-amplitude cervical manipulation targeted at C1-C2 (condition 3). Conditions 1 and 2 will be held for 1 minute before returning to neutral alignment. For the manipulation, the head will be repositioned at neutrality immediate. An experienced practitioner will perform the manipulation on the adjustable and pivotal MRI bed. After each condition, MRI of the upper neck and cerebrum for perfusion and blood flow will ensue.
Arm/Group | Intervention Group
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 20

OUTCOME MEASURES:

1. Primary Outcome: Changes in Blood Flow Through the Vertebral Artery and Posterior Cerebral and Cerebellar Circulation
Description: Phase contrast MRI provides velocity measurements that can be used for analysis of the blood flow and tissue motion. At the level of C1-2, the contralateral and ipsilateral vertebral arteries (VA), defined to the direction of head motion, were assessed and anatomical images were established to localize the VA circulation. Mean and SDs were calculated for VA blood velocity (cm/s) for each of the head conditions and VA side. Differences between task maneuvers and VA flow and velocity were evaluated using a repeated-measures analysis of variance with factors of head position and VA side, and a level of significance was set at .05
Time Frame: The series of fMRI sequences will be performed on each participant immediately after each condition. Through study completion, data will be presented after an average of 1 year.
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Intervention Group
Number analyzed (Participants) | 20
cm/s
  Neutral head position | 15.5 (3.5)
  Maximum head rotation | 15.1 (3.9)
  Cervical manipulation | 14.7 (3.6)

2. Secondary Outcome: Changes in Tissue Perfusion in the Posterior Cerebrum and Cerebellum Will be Assessed Using Arterial Spin Labeling (ASL) MRI Technique.
Description: ASL allows one to separate the blood flow from the BOLD effect, thus giving clear measures of perfusion. More specifically ASL will be used to measure blood perfusion and allow extraction of metabolic difference from flow differences in BOLD imaging. It is a quantitative technique, yielding values with units of ml/(100g of tissue)·min-1.
Time Frame: The series of ASL sequences will be performed on each participant immediately after each condition. Through study completion, data will be presented after an average of 1 year.
Measure: Mean (Standard Deviation); unit: ml/100g of tissue/minute
Groups:
- Intervention Group: Participants included in the experimental arm will be adults aged 18 years and older with chronic neck pain who have been prescribed cervical manipulation for treatment of their condition. Each participant will undergo three separate test maneuvers. Each participant will begin with neutral cervical spine as a standard natural control, followed by block randomization between maximum voluntary rotation of the cervical spine and one cervical manipulation. Please see Intervention section for a detailed description.
  Head positions and spinal manipulation: Each participant will undergo three separate test maneuvers. Neutral (0° rotation) neck position (condition 1) will be followed by block randomization between maximum voluntary rotation (condition 2) and a high-velocity-low-amplitude cervical manipulation targeted at C1-C2 (condition 3). Conditions 1 and 2 will be held fo
Arm/Group | Intervention Group
Number analyzed (Participants) | 20
ml/100g of tissue/minute
  Neutral head position | 79.2 (25)
  Maximum head rotation | 79 (25.5)
  Cervical manipulation | 80.1 (26.6)

3. Other Pre Specified Outcome: Changes in Blood Flow Through Vertebral Artery
Description: Phase contrast MRI provides velocity measurements that can be used for analysis of the blood flow and tissue motion. At the level of C1-2, the contralateral and ipsilateral vertebral arteries (VA), defined to the direction of head motion, were assessed and anatomical images were established to localize the VA circulation. Mean and SDs were calculated for VA blood flow (mL/s) for each of the head conditions and VA side. Differences between task maneuvers and VA flow and velocity were evaluated using a repeated-measures analysis of variance with factors of head position and VA side, and a level of significance was set at .05
Time Frame: The series of fMRI sequences will be performed on each participant immediately after each procedure.
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Intervention Group
Number analyzed (Participants) | 20
mL/s
  Neutral neck position | 1.8 (0.7)
  Manipulation | 1.8 (0.8)
  Maximum rotation | 1.7 (0.6)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Intervention Group: Participants included in the experimental arm will be adults aged 18 years and older with chronic/recurrent neck pain Grade II who have been prescribed cervical manipulation for treatment of their condition. Head positions and spinal manipulation: Each participant will undergo three separate test maneuvers. Neutral (0° rotation) neck position (condition 1) will be followed by block randomization between maximum voluntary rotation (condition 2) and a high-velocity-low-amplitude cervical manipulation targeted at C1-C2 (condition 3). Conditions 1 and 2 will be held for 1 minute before returning to neutral alignment. For the manipulation, the head will be repositioned at neutrality immediate. An experienced practitioner will perform the manipulation on the adjustable and pivotal MRI bed. After each condition, MRI of the upper neck and cerebrum for perfusion and blood flow will ensue.
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=20)
Minor aggravation of neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) — One patient reported minor aggravation of local neck pain. Attributed to lying on MRI table for prolonged period. Pain no longer present at follow-up 24 hours later.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT02667821/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT02667821/ICF_001.pdf